CLINICAL TRIAL: NCT06592729
Title: The Effect of Scenario-Based Simulation Method on Developing Senior Nursing Students Managerial Conflict Resolution and Problem-Solving Skills
Brief Title: Simulations Impact on Nursing Students Conflict Resolution and Problem-Solving Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Miray Aksu, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBU-HEM-MA-02
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Simulation; Training
Keywords: Scenario Based Simulation; Nursing Education
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This research will be conducted as an experimental study with pretest- posttest randomised control group design
Who Masked: Participant
Masking Description: Experimental and control groups will be determined using https://www.randomizer.org
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conflict and problem solving scenario training (Experimental groups) (Experimental): The experimental group will be taken to scenario-based simulation. The simulation application will be taken to the case suitable for the conflict resolution skills and problem solving skills of the final year students. Before the simulation, students will be informed about the scenario (prebriefing) and expectations will be shared. This stage will take approximately 10 minutes. The student will be given time to solve the conflict for 15 minutes. At the end of the scenario, the student will be taken to the debriefing session.
  Interventions: Behavioral: education
- conflict and problem solving curriculum training (Control groups9 (No Intervention): Control group students will take 8 hours of theoretical courses on Conflict Resolution (4 hours) and Problem Solving (4 hours).

INTERVENTIONS:
Behavioral: education — intervention group was taken to scenario-based simulat
  Arms: conflict and problem solving scenario training (Experimental groups)

SUMMARY:
Scenario-based simulation training effectively enhances nursing students' core competencies, communication, teamwork, problem-solving, and decision-making skills, better preparing them for real-world experiences. This research focuses on the impact of scenario-based simulations in developing conflict resolution and problem-solving skills in nursing management courses. By imitating real-life clinical scenarios, such training can improve students' abilities to manage conflicts and address clinical challenges, making them more effective and competent in clinical settings after graduation. The study aims to provide educators with insights and practical recommendations for incorporating innovative methods into nursing education programs.

DETAILED DESCRIPTION:
Scenario-based simulation training is highly effective in developing nursing students' core competencies, clinical skills, teamwork, problem-solving, and decision-making abilities. This training provides a safe and supportive environment for students to practice and develop the communication skills necessary for nursing practice, helping them prepare better for real-world experiences and increasing their confidence and sensitivity in complex situations. It has also been shown to enhance students' interest in learning and participation because it improves their ability to understand and apply teaching content. Based on these studies, it is important to incorporate scenario-based simulation training into nursing education programs to further develop students' competencies.

Scenario-based simulations stand out as an effective learning tool by offering students learning environments that mimic real-world scenarios, allowing them to gain experience. Scenario-based simulation training gives students the opportunity to experience realistic situations they may encounter in clinical settings, apply theoretical knowledge in practice, develop effective communication, collaboration, and teamwork skills, learn from their mistakes and successes, and increase their confidence. Considering all this information, using scenario-based simulation training in nursing management courses can help students develop conflict resolution and problem-solving skills in nursing management by imitating real-life clinical scenarios, providing them with an interactive learning environment that will help them work more effectively and competently in clinical settings after graduation.

Preparing nursing students for the clinical environment and the rapidly changing business world makes it important to develop conflict resolution and problem-solving skills before graduation. Conflict resolution and problem-solving skills are among the basic requirements for successfully operating in the modern business world. Conflict resolution techniques, such as mediation, negotiation, and compromise, help students manage conflicts between members of the clinical care team, patients, and their families. Additionally, problem-solving skills enable students to identify and address clinical challenges, enhancing their ability to provide quality healthcare. By developing these skills, nursing students can increase their adaptation to and satisfaction with clinical practice. Problem-solving skills are positively influenced by positive attitudes towards communication and seeing oneself as an initiator. Therefore, having conflict resolution and problem-solving skills can positively impact students' future professional and social success, playing a significant role in making them more effective and efficient in their work life. Some studies in the literature suggest that there is a relationship between nursing students' problem-solving skills and conflict resolution skills; when students' problem-solving skills are high, their conflict resolution skills may also increase. This hypothesis suggests that students' cognitive abilities and problem-solving strategies can be more effective in coping with various situations and in conflict resolution processes.

This research aims to determine the effect of scenario-based simulation methods in developing managerial conflict resolution and problem-solving skills in pre-graduation students. The theoretical framework of the research will consist of literature covering learning theories, management education in nursing, and the use of simulation in curricula to provide a deeper understanding and interpretation of the research findings. It is believed that this research will provide significant information for educators and educational policymakers in improving learning environments and developing effective strategies for students to enhance their essential skills. In addition to forming practical recommendations for making educational processes more effective, it is thought that the design and implementation of programs using innovative methods in education will demonstrate the impact on the skill development of pre-graduation nursing students. These contributions can enhance nursing management course curricula and help students successfully take on leadership roles and positions in society in the near future.

ELIGIBILITY:
Inclusion Criteria:

* To be a senior student at Gülhane Faculty of Nursing,
* Students' voluntary acceptance to participate in the research,
* To have taken the conflict management and problem solving course for the first time,

Exclusion Criteria:

* To have received training on conflict management and problem solving outside the course,
* Failure to complete any of the measurement tools

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Conflict Action Styles Scale | four weeks
  The scale is five-point Likert type and consists of 35 items and 5 sub-factors. The sub-factors of the scale consist of avoidant (statements 1, 6, 11, 16, 21, 26 and 31), coercive (statements 2, 7, 12, 17, 22, 27 and 32), facilitative (statements 3, 8, 13, 18, 23, 28 and 33), conciliatory (statements 4, 9, 14, 19, 24, 29 and 34) and confrontational (statements 5, 10, 15, 20, 25, 30 and 35). In which sub-dimension the highest score is obtained, that sub-dimension determines the conflict action style of the person.

SECONDARY OUTCOMES:
Problem Solving Inventory | four weeks
  The inventory is a Likert-type scale consisting of 35 items scored between 1-6. According to this inventory, the lowest score is 32 and the highest score is 192. High total scores indicate that the individual perceives himself/herself as inadequate in problem solving skills, while low scores indicate effectiveness in problem solving and behaviours and attitudes related to successful problem solving.

CONTACTS AND LOCATIONS:
Overall Officials: Miray Aksu, Phd, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No